CLINICAL TRIAL: NCT06317896
Title: Value of Dynamic Monitoring of Early Recurrence of Hepatocellular Carcinoma After Radical Resection Based on CTCS: a Prospective Cohort Study
Brief Title: Value of Dynamic Monitoring of Early Recurrence of Hepatocellular Carcinoma After Radical Resection Based on CTCS
Status: Not yet recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-KY-048-01
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Hepatocellular Carcinoma; Circulating Tumor Cell; Recurrence; Surgery
Keywords: Hepatocellular Carcinoma; Circulating Tumor Cell; Recurrence; Dynamic Monitoring
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplastic Cells, Circulating; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with hepatocellular carcinoma: Patient with hepatocellular carcinoma who can undergo radical resection
  Interventions: Diagnostic Test: circulating tumor cells

INTERVENTIONS:
Diagnostic Test: circulating tumor cells — blood sample and tissue specimen for circulating tumor cell and DNA will be done to patient with hepatocellular carcinoma
  Other Names: circulating tumor cell DNA

SUMMARY:
On the basis of previous retrospective studies, the Task Force will further optimize the CTCs longitudinal surveillance model and initially validate the subclonal origin (CTC-DNA) of recurrent/metastatic foci derived from CTCs at the molecular level in hepatocellular carcinoma, prospective clinical trials will be conducted to further validate the predictive value of the CTCS longitudinal monitoring model in predicting postoperative recurrence of hepatocellular carcinoma, and to verify whether it is earlier than imaging to indicate recurrence, to explore the clinical feasibility of CTCs in guiding postoperative adjuvant therapy of liver cancer, and to provide new ideas for early intervention strategy of liver cancer after operation, to establish a set of standardized clinical scheme of auxiliary treatment for patients with liver cancer after operation for accurate and individualized"Early diagnosis and treatment".

DETAILED DESCRIPTION:
The recurrence rate of HCC after radical resection is high. MRD is the root cause of HCC recurrence, and the MRD result is an important basis for auxiliary treatment decision-making after radical resection. On the basis of previous retrospective studies, the Task Force will further optimize the CTCs longitudinal surveillance model and initially validate the subclonal origin (CTC-DNA) of recurrent/metastatic foci derived from CTCs at the molecular level in hepatocellular carcinoma, prospective clinical trials will be conducted to further validate the predictive value of the CTCS longitudinal monitoring model in predicting postoperative recurrence of hepatocellular carcinoma, and to verify whether it is earlier than imaging to indicate recurrence, to explore the clinical feasibility of CTCs in guiding postoperative adjuvant therapy of liver cancer, and to provide new ideas for early intervention strategy of liver cancer after operation, to establish a set of standardized clinical scheme of auxiliary treatment for patients with liver cancer after operation for accurate and individualized"Early diagnosis and treatment", to provide high-quality evidence-based medicine for the clinical practice of preventing recurrence after radical hepatectomy

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18-75 years;
2. Preoperative imaging examination diagnosed hepatocellular carcinoma (BCLC) stage 0 /stage A/stage B, eligible for radical surgery;
3. ECOG physical status score is 0-1;
4. Child-Pugh score is 5-6 points (Level A);
5. Not received any anti-tumor therapy;
6. Laboratory tests were at normal levels within 7 days before enrollment.

Exclusion Criteria:

1. Patient can't provide blood samples for CTCs and CTC-DNA testing;
2. Patient with two or more types of tumors at the same time;
3. Non-primary liver lesions;
4. Pregnant or lactating women;
5. Patient with a history of other malignant tumors within the past 5 years or at the same time, except cured skin basal cell carcinoma, cervical carcinoma in situ and thyroid papillary carcinoma;
6. Patient with serious heart disease;
7. Other conditions deemed unsuitable for inclusion by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with hepatocellular carcinoma who can undergo radical surgical resection
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence-free survival rate | 2 years
  percentage of recurrence-free survival 2 years after surgery

SECONDARY OUTCOMES:
Correlation between CTCs status dynamic changes and relapse | 2 years
  Correlation between CTCs status dynamic changes and relapse
Correlation between metastasis，primary tumor and CTCs in blood through NGS and CTC-DNA | 2 years
  The subclonal origin of recurrent/metastatic foci derived from CTCs was verified at the molecular level in hepatocellular carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Mingxin Pan, Prof., Principal Investigator — Southern Medical University, China
Locations (3):
- China (3):
  - The Sixth Affiliated Hospital of South China University of Technology, Foshan, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou, Guangdong